CLINICAL TRIAL: NCT04897633
Title: Modulation of Cognitive Control Via Transcranial Continuous Electrical Stimulation of Additional Motor Areas in Parkinson's Patients
Acronym: STAR-PARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-46; ID-RCB (Other: 2020-A03170-39)
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: transcranial stimulation; tDCS; simon task
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients ON (Experimental): Patients will performed Simon's task with tDCS active or sham when treatment is OFF (for standard care procedure)
  Interventions: Device: transcranial electric stimulation
- Patients OFF (Experimental): Patients will performed Simon's task with tDCS active or sham when treatment is ON (for standard care procedure)
  Interventions: Device: transcranial electric stimulation
- Healthy volunteers (Experimental): Healthy volunteers will performed Simon's task with tDCS active or sham
  Interventions: Device: transcranial electric stimulation

INTERVENTIONS:
Device: transcranial electric stimulation — Simon's task assessment when under tDCS
  Other Names: DC STIMULATOR PLUS

SUMMARY:
In Parkinson's disease (PD), recent work has shown that dopaminergic treatments alter one of the two aspects of impulsivity: they do not alter the propensity to produce "automatic" responses, but deteriorate the ability to inhibit and correct (that is, control) them. In healthy subjects, the investigator's team has also demonstrated that transcranial direct current "cathodal" electrical stimulation (tDCS) of Supplementary Motor Areas decreases the frequency of behavioral errors by improving the ability to "correct" responses.

The main objective of this project is to determine whether cathodal tDCS of Supplementary Motor Areas in PD patients under dopaminergic treatment improves the control and correction of errors about to be made and compensates for the deficits induced by the treatment.

All participants will perform a reaction time task of choice (Simon's task), with and without ("sham" session) tDCS. The experimental design of this single-center, single-blind, randomized study will be that of 3 parallel groups (treated Parkinson's disease, untreated Parkinson's disease patient, and matched control subjects) with cross-over application of tDCS. All participants will be blind to the operating mode of the tDCS (either functional or in "sham" mode corresponding to a control condition). The order of the sessions (with and without tDCS) will be randomized within each of the 3 groups of subjects. The analysis of errors about to be made but inhibited in time (known as "early errors") will be carried out through electromyographic (surface) recording of muscle activities involved in motor responses.

tDCS is expected to improve the ability of treated patients to correct their errors about to be made. This study will thus provide a better understanding of the mechanisms of action control and possibly propose a new therapeutic approach for treatment-induced impulsivity disorders in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria for Parkinsonien patients:

* Age> 18 years old
* Idiopathic Parkinson's disease meeting the diagnostic criteria as defined by Ward and Gibb (1990)
* Patients usually taking dopaminergic treatment.
* No cognitive deterioration with: a Montreal Cognitive Assessment (MoCA) score ≥ 26
* Patient with Parkinson's disease in the advanced motor complications stage for which surgical treatment is being considered

Inclusion Criteria for healthy subjects

* Age> = 18 years old
* Patient free from Idiopathic Parkinson's Disease
* No cognitive deterioration: MMSE (MiniMentalSate Evaluation)> 26

Exclusion Criteria for both parkinsonien patients an healthy volunteers:

* Uncorrected altered visual acuity
* Dyschromatopsia (especially color blindness)
* Psychotropic treatment introduced or modified recently (<1 month)
* Wearing a pacemaker (Pace Maker or Implantable Defibrillator)
* Pregnancy (verified by a urine pregnancy test for women of childbearing age)
* Other central nervous system disease (other parkinsonian syndrome, epilesia, stroke, etc.) or peripheral
* Intracranial metal implants on the cephalic stage and cochlear implant
* Untreated progressive mood or psycho-behavioral disorder
* Severe and poorly controlled eczema

Exclusion criteria for Parkinson's patients only:

* Significant and disabling abnormal movement, not allowing good acquisition of the EMG signal (tremors or dyskinesias)
* Wearer of a Deep Brain Stimulation device (CI at tDCS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Rapid error rate. | Day 2
  Responses recorded on the opposite side to that expected
Rapid error rate. | Day 3
  Responses recorded on the opposite side to that expected

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier ARNAUD, Study Director — APHM
Locations (1):
- Service Neurologie et pathologies du mouvement, Marseille, France

IPD SHARING:
Plan to Share IPD: No